CLINICAL TRIAL: NCT04337034
Title: Participation in Everyday Life - A Randomized Controlled Trial of Mobile Phone-supported and Family-centred Rehabilitation After Stroke in Uganda.
Brief Title: F@ce 2.0 a Mobile Phone-supported and Family-centred Rehabilitation Intervention After Stroke in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Susanne Guidetti, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: F@ce 2.0
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to participate in F@ce 2.0 (IG) or a control group (CG) receiving usual rehabilitation at two different sites; both an urban (IG+CG) and rural site (CG+IG) in Uganda
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mobile phone supported and family-centred rehabilitation (Experimental): Participants in the intervention group will receive an 8-week mobile phone supported and family-centred rehabilitation intervention (F@ce 2.0)
  Interventions: Behavioral: Mobile phone supported and family-centred rehabilitation; Procedure: Information and blood pressure measurement
- Information and blood pressure measurement (Active Comparator): Control group participants will be given information about stroke and their blood pressure will be measured
  Interventions: Procedure: Information and blood pressure measurement

INTERVENTIONS:
Behavioral: Mobile phone supported and family-centred rehabilitation — Participants in the intervention group will receive an eight-week mobile phone supported and family-centred rehabilitation intervention (F@ce 2.0).The participants will be introduced to a problem-solving strategy intended to facilitate the learning and problem-solving process to be used during the intervention. The strategy will provide a structure for healthcare professionals delivering the intervention. Three targets (goals) in daily activities will be formulated that the person wants and needs to do within the home environment. Each activity will be practiced together with the healthcare professionals and family members. Family members will be informed about the participant's target activities and the planned strategies for reaching the targets. The participants will practice the target activities in their home environment supported by mobile phone calls and SMS. In addition they will be given information about stroke and their blood pressure will be measured.
  Arms: mobile phone supported and family-centred rehabilitation
Procedure: Information and blood pressure measurement — Control group participants will be given information about stroke and their blood pressure will be measured.

SUMMARY:
The purpose of the present proposal is to implement and evaluate a new model for mobile phone supported and family-centred rehabilitation intervention (F@ce 2.0) with regard to functioning in activities in daily living and participation in everyday life among persons with stroke and their families (in rural and urban areas) in Uganda.

DETAILED DESCRIPTION:
The investigators' previous feasibility study suggested beneficial effects on self-efficacy and occupational performance and satisfaction of a mobile phone supported and family-centred rehabilitation intervention (F@ce1.0) after stroke in Uganda. The purpose of the present proposal is to implement and evaluate F@ce on functioning in activities in daily living (ADL) and participation in everyday life among persons with stroke and their families.

With recommendations on evaluation of complex interventions both outcomes and processes will be studied and hence both quantitative and qualitative methods will be applied. In a randomized controlled trial F@ce 2.0 will be evaluated compared to ordinary rehabilitation in urban/rural Uganda regarding; self-efficacy, perceived performance and participation in everyday activities, independence in ADL, health care utilization and the families´ perceived participation in everyday activities. Qualitative data will explore experiences of people with stroke and family members of participating in F@ce 2.0. This research program has a multidisciplinary perspective for sustainable rehabilitation, a prerequisite for better living conditions for people with stroke in low/middle income countries.

ELIGIBILITY:
Inclusion Criteria:

* stroke diagnosis identified with CT scan or clinical symptoms
* inhabitant in a rural part of Kalungu District, near Masaka Uganda, or Kampala with surroundings
* access to and ability to use a mobile phone
* ability to speak and express themselves in English and/or Luganda
* Modified Rankin Scale level 2 to 4.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Self-efficacy Scale | Differences in change between baseline and 3, 6 and 12 months
  Participants are instructed to rate how confident they feel about performing each of 16 everyday activities on a 10-point rating scale ranging from 1) "not confident at all in my ability" to 10) "very confident in my ability". The average of all responses are calculated.

SECONDARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | Differences in change between baseline and 3, 6 and 12 months
  COPM measures performance and satisfaction in self-care, productivity and leisure from the individual's perspective using a scale of 1-10. The participant is asked 1) to rate performance of the specified activities using a 1 to 10 scale and 2) to score his or her satisfaction with that performance using the same scale. Weighted scores of the chosen activities are added separately for performance and satisfaction to create two summative scores. The summative scores are then divided by the number of rated activities to provide COPM scores.
Stroke Impact Scale (SIS) 3.0 Uganda version | Differences in change between baseline and 3, 6 and 12 months
  Assesses the perceived impact on functioning in everyday life in eight domains: Strength, Memory and thinking, Emotions, Communication, ADL/ Instrumental activities of daily living (IADL), Mobility, Hand function and Participation. The SIS includes 59 items within these eight domains. Aggregated scores ranges from 0 to 100, the higher the score, the lower the perceived impact of stroke, i.e. fewer problems in everyday life. The SIS 3.0 also includes a question to assess the participant's global perception of recovery presented in a vertical analogue scale ranging from '0 = no recovery to 100 = full recovery'.
Barthel Index | Differences in change between baseline and 3, 6 and 12 months
  Measures independence in 10 self-care and mobility activities. Scores range from 0 to 100, with a lower score indicating greater dependency.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Guidetti, Professor, Principal Investigator — Karolinska Institutet
Locations (3):
- Uganda (3):
  - Mulago Hospital, Kampala
  - Stroke Rehabilitation Centre, Kampala
  - Masaka Hospital, Masaka

IPD SHARING:
Plan to Share IPD: No